CLINICAL TRIAL: NCT03216603
Title: Health Literacy. An Intervention on Organized Information and Health Care for People With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Health Literacy in People With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian Extra Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Christine Råheim Borge, Researcher, Lovisenberg Diakonale Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 298
Record Dates: First submitted 2017-07-07; First posted 2017-07-13 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Health literacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health literacy intervention group (Experimental): Health literacy intervention group will receive self-management help using a motivating interviewing technique delivered by nurses trained on motivating interviewing technique and COPD.
  Interventions: Behavioral: Health literacy intervention group
- Usual care group (No Intervention): Usual care group will receive usual follow up

INTERVENTIONS:
Behavioral: Health literacy intervention group — In the health literacy intervention group all patients will receive self-management help using a motivating interviewing (MI) technique delivered by two MI and COPD trained nurses once a week for eight weeks after hospitalization. Subsequently, the contact between the patients and the nurses will be by follow up motivational telephone calls once a month or more if needed for four months (i.a a total of six months intervention period).
  Arms: Health literacy intervention group

SUMMARY:
Health literacy refers to personal and relational factors affecting a person's ability to acquire, understand and use information about health and health services. In a need assessment study it was found that, the health services need to focus on health literacy factors in the follow up of patients with chronic obstructive pulmonary disease (COPD).

Thus, this project evaluate the effect a of a health literacy partnership health promotion intervention (hospital, municipalities, university) after discharge from hospital with the use of motivational interviewing and tailored follow-ups on re-admission, health literacy, self-management quality of life and cost in people with COPD compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD,
* Above 18 years,
* Admitted to a medical department at the main intervention hospital, l
* Live in the sites belonging to the intervention hospital.

Exclusion Criteria:

* Not diagnosed with COPD,
* Not above 18 years,
* Not admitted to a medical department at the main intervention hospital, and
* Not living in the sites belonging to the intervention hospital.
* Cognitive failure
* Patients that are investigated or treated for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of admissions | Eight weeks, six months and one year
  Number of re-admissions

SECONDARY OUTCOMES:
Change of health literacy | Eight weeks, six months and one year
  Questionnaire
Change of disease specific quality of life | Eight weeks, six months and one year
  Questionnaire
Change of e-Health | Eight weeks, six months and one year
  Questionnaire
Change of physical function | Eight weeks, six months and one year
  Questionnaire
Change of self-management | Eight weeks, six months and one year
  Questionnaire
Change of psychological stress | Eight weeks, six months and one year
  Questionnaire
Change of self-efficacy | Eight weeks, six months and one year
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christine Borge, Phd, Principal Investigator — University of Oslo and Lovisenberg Diaconal Hospital; Astrid K. Wahl, Phd, Study Chair — University of Oslo
Locations (1):
- Lovisenberg Diakonale Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen MH, Wahl AK, Borge CR. Patients' and healthcare personnel's experiences of a health-literacy intervention in chronic obstructive pulmonary disease - a qualitative study. BMC Health Serv Res. 2025 Sep 30;25(1):1256. doi: 10.1186/s12913-025-13299-z. PMID 41029694
- [Derived] Borge CR, Larsen MH, Osborne RH, Aas E, Kolle IT, Reinertsen R, Lein MP, Thorn M, Lind RM, Groth M, Strand O, Andersen MH, Moum T, Engebretsen E, Wahl AK. Impacts of a health literacy-informed intervention in people with chronic obstructive pulmonary disease (COPD) on hospitalization, health literacy, self-management, quality of life, and health costs - A randomized controlled trial. Patient Educ Couns. 2024 Jun;123:108220. doi: 10.1016/j.pec.2024.108220. Epub 2024 Feb 16. PMID 38458089